CLINICAL TRIAL: NCT01547845
Title: The NCl Community Cancer Center Program Patients Reported Symptom Surveillance and Disparities Study
Brief Title: Cancer Symptom Data From Multiple Treatment Centers
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999912039; 12-C-N039
Record Dates: First submitted 2012-03-06; First posted 2012-03-08 (Estimated); Last update posted 2019-05-28 (Actual); Status verified 2019-05-23

CONDITIONS: Breast Cancer; Colon Cancer
Keywords: Disparities; Patient Reported Outcomes; Symptoms; Symptom Surveillance
MeSH Terms: conditions — Breast Neoplasms; Colonic Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

SUMMARY:
Background:

- Cancer and cancer treatments can cause symptoms and side effects. Pain, fatigue, and emotional distress are three common symptoms. Accurate reporting of these symptoms can improve treatment methods and outcomes. Even though symptom reporting is important to treatment, there is no method to collect and compare patient data from multiple cancer care centers. Researchers want to develop a method for collecting cancer patient symptom information from multiple centers. This method may help improve cancer treatment at hospitals and other care centers.

Objectives:

- To collect patient-reported symptom information from multiple cancer care centers.

Eligibility:

* Individuals at least 21 years of age who were treated for breast or colon cancer in the past year.
* Participants will come from one of the participating cancer care centers.

Design:

* Participants will answer a short questionnaire about their symptoms during cancer treatment. Questions will ask about symptom severity and experiences. Other questions will ask how well the doctors and nurses managed the symptoms.
* Participant responses will be compared with other medical and personal information. This information may include cancer type, age at diagnosis, and type of treatment.
* Treatment will not be provided as part of this study.

DETAILED DESCRIPTION:
Background:

* Cancer and its treatment lead to symptoms and side effects. Pain, fatigue, and emotional distress are three of the most common and distressing symptoms. Patient report is the gold standard for assessing these symptoms and is critical to patient-centered care.
* Symptoms are often under-reported or under-treated leading to impairments in quality of life, functioning, and treatment adherence. Factors contributing to under-reporting/treatment occur within patients (e.g., fear of addiction to pain meds), providers (e.g., lack of training), and the healthcare system (e.g., under-insurance).
* A limited number of studies suggest that the burden symptoms falls unevenly on certain racial/ethnic, socioeconomic status (SES), and insurance status groups.
* Despite the importance of symptoms in cancer care, there is no method for systematically collecting patient reported data at institutional or national levels. Such a system could identify at risk groups, inform intervention, and ultimately improve quality of care.
* This study uses existing resources to design a cost-effective symptom surveillance system. The NCI Community Cancer Center Program (NCCCP) provides the infrastructure for efficiently conducting a multi-site pilot in a real-world setting with a diverse sample of patients. The Commission on Cancer s Rapid Quality Reporting System (RQRS) will automate sampling to minimize burden on the cancer center s staff, facilitate data collection during or soon after treatment, and protect patients personal identifiers. The survey instrument is based upon previously validated measures.

Objectives:

* To pilot a method for collecting patient reports of symptom-related experiences that could be used for surveillance at institutional and, in the future, population levels.
* To investigate disparities in symptom burden and management between racial/ethnic, SES, and health insurance status groups.
* To pilot the use of patient-reported symptom data for quality improvement of symptom management at participating cancer centers.

Eligibility:

* Diagnosed with Stage I-III breast or colon cancer as first primary cancer between February 2011 and January 2013
* Age of 21 years or older
* Received cancer care from one of 17 participating NCCCP Cancer Centers.

Design:

* This cross-sectional survey will collect reports of symptoms and related experiences from patients 3-12 months after cancer diagnosis via mailed questionnaire. A methodological experiment will randomize patients after the second mailing to compare telephone follow-up to a third mailing. Data on cost and Cancer Center staff time will be collected to provide scalable estimates of overall cost and examine cost-effectiveness of telephone follow-up.
* The study will provide prevalence estimates for various symptoms and symptom management items. More complex, model-based statistics will be used to investigate symptom disparities (Aim 2). For these models, outcomes will be either continuous (e.g., pain severity) or ordinal (e.g., symptom management items) and will be analyzed using Generalized Linear Mixed Models (GLMM) to take into account the two-level structure of the data (patients nested within Cancer Centers). We expect to enroll 2,550 patients.

ELIGIBILITY:
* INCLUSION CRITERIA:

The respondent universe will consist of all cancer patients at the 16 participating NCCCP Cancer Centers who satisfy the following conditions:

* Diagnosed with Stage I-III breast or colon cancer as first primary cancer between February 2011 and January 2013
* Eligible for one of the RQRS breast or colon Quality of Care Indicators
* Age of 21 or older
* Not known to be deceased at the time of contact

The NCCCP is a network of 30 community hospitals in 22 states supporting cancer research and enhancing cancer care for patients close to home. Most cancer patients in the U.S. are diagnosed and treated at community hospitals; not in NCI Comprehensive Cancer Centers where much research is conducted. The National Cancer Institute Community Cancer Centers Program (NCCCP) is expanding cancer research and bringing advanced cancer treatments to patients in community hospitals in rural, suburban and inner-city areas.

This study is being conducted at the 16 pilot NCCCP sites that first entered the program in 2007. All 16 participate in RQRS. These 16 pilot sites are located in 14 states throughout the United States.

EXCLUSION CRITERIA:

* Patients will be excluded for the following reasons:Patient is ineligible for one of the 5 RQRS breast or colon quality indicators
* Patient is deceased at the time of sampling
* Patient has Stage IV cancer

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2517 (Actual)
Dates: Start 2012-02-10; Study Completion 2019-05-23

PRIMARY OUTCOMES:
PRO symptom measurement | 4-9 months post treatment
  Complete reporting of symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Castro, R.N., Principal Investigator — National Cancer Institute (NCI)
Locations (15):
- United States (15):
  - St. Joseph's Orange, Orange, California
  - Penrose Cancer Center, Colorado Springs, Colorado
  - Hartford Hospital, Hartford, Connecticut
  - Christiana Care Health Services, Newark, Delaware
  - Northside Hospital, Atlanta, Georgia
  - St. Joseph's/Candler Health System, Savannah, Georgia
  - Our Lady of the Lake/ Mary Bird Perkins, Baton Rouge, Louisiana
  - The Cancer Institute Catholic Health Initiatives, Towson, Maryland
  - Billings Clinical Cancer Center, Billings, Montana
  - CHI, St. Fancis, Grand Island, Nebraska
  - CHI, Good Samaritan, Kearney, Nebraska
  - Lehigh Valley Hospital, Allentown, Pennsylvania
  - Spartanburg Regional Hospital, Spartanburg, South Carolina
  - Sanford Health, Sioux Falls, South Dakota
  - Ascension Health Systems, Milwaukee, Wisconsin

REFERENCES:
- [Background] Arora NK, Reeve BB, Hays RD, Clauser SB, Oakley-Girvan I. Assessment of quality of cancer-related follow-up care from the cancer survivor's perspective. J Clin Oncol. 2011 Apr 1;29(10):1280-9. doi: 10.1200/JCO.2010.32.1554. Epub 2011 Feb 28. PMID 21357781
- [Background] Banna GL, Collova E, Gebbia V, Lipari H, Giuffrida P, Cavallaro S, Condorelli R, Buscarino C, Tralongo P, Ferrau F. Anticancer oral therapy: emerging related issues. Cancer Treat Rev. 2010 Dec;36(8):595-605. doi: 10.1016/j.ctrv.2010.04.005. Epub 2010 Jun 8. PMID 20570443
- [Background] Anderson KO, Green CR, Payne R. Racial and ethnic disparities in pain: causes and consequences of unequal care. J Pain. 2009 Dec;10(12):1187-204. doi: 10.1016/j.jpain.2009.10.002. PMID 19944378